CLINICAL TRIAL: NCT02255188
Title: Evaluate Hemocompatibility Vascular Prosthesis to Prevent Its Thrombosis
Brief Title: Experimental Study of the Vascular Prosthesis Manufactured by Electrospinning
Status: Completed | Type: Observational
Sponsor: Meshalkin Research Institute of Pathology of Circulation (Network)
Responsible Party: Sponsor
Other Study IDs: 16.01.2014 № 2
Record Dates: First submitted 2014-09-10; First posted 2014-10-02 (Estimated); Last update posted 2017-09-08 (Actual); Status verified 2015-07

CONDITIONS: ARTERIAL OCCLUSIVE DISEASE
Keywords: Haemostas, prosthesis
MeSH Terms: conditions — Arterial Occlusive Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (4):
- Graft type - PCL: PCL - polycaprolactone
  Interventions: Procedure: blood sampling procedure
- Graft type - PCL/ gelatin: polycaprolactone/ gelatin/poorly permeable layer;
  Interventions: Procedure: blood sampling procedure
- Graft type - PLGA/PCL/gelatin: PLGA/PCL/gelatin - polylactide-co-glycolide / polycaprolactone / gelatin/poorly permeable layer
  Interventions: Procedure: blood sampling procedure
- Graft type - nylon 6
  Interventions: Procedure: blood sampling procedure

INTERVENTIONS:
Procedure: blood sampling procedure — 30 ml of venous blood will be collected from all voluteers using a special vacuum tubes after informed consent. Blood sampling is carried out from an arm vein. All subsequent studies will be executed in the laboratory diagnostic division of Novosibirsk Research Institute of Circulation Pathology and the presence of the donors is unnecessary

SUMMARY:
The purpose of this study is to determine whether the Vascular prosthesis manufactured by Electrospinning is safe with respect to the development of thrombosis.

DETAILED DESCRIPTION:
To test the influence of the prostheses to hemostasis blood will be pumped through the vascular prosthesis or control silicone tube (both with identical inner diameter 1,7 mm) during 20 minutes at a linear velocity 10 cm/sec (corresponding to 18 ml/min). The tested prostheses (or control tubes) will be installed between two syringes with blood installed in the UTPS-1 instrument providing synchronical movement of pistons of both syringes. Installing UTPS-1 was designed and manufactured at the Institute of Chemical Biology and Fundamental Medicine, Siberian Branch of the Russian Academy of Sciences consists of a mechanical pushers, equipped with clamps for syringes and pistons, stepper motor, electronic control unit and power supply.

UTPS-1 and polypropylene non-pyrogenic syringes filled with blood without any bulbs of air provides absence of contacts with air, pyrogens and minimize lysis of blood cells. UTPS-1 has no analogues, and does not require licensure, metrological control or obtaining of any other permits.

After pumping the blood will be separated into plasma and cell fraction according to standard laboratory methods. Primary blood (before any treatment), blood after pumping through silicon tube (control), and vascular prosthesis will be tested for hemostatic parameters.

Notification of basic and additional parameters being studied, which will be

evaluated in the study:

1. The initial parameters of blood hemostasis will be evaluated (Platelet count; Platelet aggregation; Prothrombin time, International Normalised Ratio [INR], activated partial thromboplastin time (aPTT), prothrombin Quick, thrombin time, soluble fibrin monomer complexes (SFMC), free hemoglobin and P- selectin concentrations).
2. To evaluate the influence of the prosthesis to circulating blood the same hemostasis characteristics wiil be evaluated in blood after 20 min of circulation through prosthesis and silicon tube (Platelet count; Platelet aggregation; Prothrombin time, International Normalised Ratio [INR], activated partial thromboplastin time (aPTT), prothrombin Quick, thrombin time, soluble fibrin monomer complexes (SFMC), the measurement of free hemoglobin, P- selectin).
3. Microscopy: a study of adhesion of blood cells on the surface of the prosthesis

Description of Design of the Research: this will be prospective (are marked in section Detailed Description)

Monocentred research

Defined indicators for each prosthesis

1. hemostasis characteristics listed hereinabove for untreated blood (control)

2 hemostasis characteristics listed hereinabove in blood after 20 min circulation through silicone tube (control)

3 hemostasis characteristics listed hereinabove in blood after 20 min circulation through After the interaction with the experimental vascular prosthesis

Will be studied 4 types of vascular prostheses made by electrospinning

* polycaprolactone;
* polycaprolactone / gelatin/poorly permeable layer;
* polylactide-co-glycolide / polycaprolactone / gelatin/poorly permeable layer;
* nylon 6

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged from 18 to 50 years at the date of the informed consent signing;
* Patients without atherosclerosis
* Patients without blood pathology

Exclusion Criteria:

* Patient did not sign the informed consent.
* Early postoperative period.
* Concomitant diseases such as atherosclerosis, blood pathology, venous thrombosis, malignancy, terminal cancer, infectious - inflammatory disease at the time of the study.
* Patients after implantation of a cardioverter-defibrillator; prior prosthetic heart valves or other implants, which can lead to mechanical damage to the blood cells.
* Receiving anticoagulants, antiplatelet, antibacterial drugs, NSAIDs.
* Myocardial infarction less than 3 months ago.
* Irreversible failure of major organs with an expected survival time of less than 1 year
* Pregnancy, lactation.
* Age above 50 years.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: volunteers, donors
Sampling Method: Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2014-10; Primary Completion 2015-10 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Number of participants (blood samples) having a higher degree of aggregation of platelets after interaction with the prosthesis, as a sign of thrombosis. (with ristomycin, adrenaline, collagen, ADP) | during the day
  percentage

SECONDARY OUTCOMES:
Platelet count | during the day
  cells / L
Prothrombin time | during the day
  seconds

OTHER OUTCOMES:
International Normalised Ratio | during the day
activated partial thromboplastin time | during the day
  seconds
prothrombin Quick | during the day
thrombin time | during the day
  seconds
soluble fibrin monomer complexes | during the day
  0-4mg/100ml
free hemoglobin | during the day
  g / l
P- selectin concentrations | during the day
  ng / ml
Adhesion of blood cells on the surface of the prosthesis | during the day
  microscopy

CONTACTS AND LOCATIONS:
Locations (1):
- popova Irina, Novosibirsk, Novosibirskay Obl., Russia